CLINICAL TRIAL: NCT00533195
Title: UVA1 Phototherapy Versus 5-MOP UVA Photochemotherapy for Patients With Severe Generalized Atopic Dermatitis
Brief Title: Comparison of UVA1 Phototherapy Versus Photochemotherapy for Patients With Severe Generalized Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Prof. Dr. Adrian Tanew, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 03/01/07; EudraCT-Nr.: 2006-00698217
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Atopic Dermatitis
Keywords: UVA1; PUVA; atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — 5-Methoxypsoralen; Methoxsalen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0 (Active Comparator): 5-MOP photochemotherapy. Intake of Geralen capsules (1.2 mg/kg) 2 hours before irradiation. Determination of the minimal phototoxic dose (MPD) and Geralen serum level prior to treatment. Start with 70 % of the MPD, no dose increments in the first treatment week. From the second week increments of the UVA dose by 20 % in the absence of an erythemal reaction, respectively by 10 % in cases of a barely perceptible erythemal response. Increments of the UVA dose at the earliest 96 hours after the last increments. Treatment frequency 3 x week for 5 weeks (=15 exposures). No maintenance therapy except emollients.
  Interventions: Drug: 5-Methoxypsoralen
- 1 (Experimental): UVA1 phototherapy. Treatment 5 x week for 3 weeks (=15 irradiations). Determination of the UVA 1 MED prior to treatment. Start with 1 MED. Increments of the UVA 1 dose in 20 % steps until a maximal dose of 70 J/cm2 in the absence of an erythemal reaction and by good tolerability. No maintenance therapy except emollients.
  Interventions: Device: UVA1 phototherapy

INTERVENTIONS:
Drug: 5-Methoxypsoralen — 1,2 mg/kg 2 hours before UVA irradiation p.o. 3 times weekly for 5 weeks
  Other Names: 5-MOP, Geralen
  Arms: 0
Device: UVA1 phototherapy — Treatment 5 x week for 3 weeks (=15 irradiations). Determination of the UVA 1 MED prior to treatment. Start with 1 MED. Increments of the UVA 1 dose in 20 % steps until a maximal dose of 70 J/cm2 in the absence of an erythemal reaction and by good tolerability.
  No maintenance therapy except emollients.
  Other Names: UVA1
  Arms: 1

SUMMARY:
The purpose of this study is to compare the efficacy, tolerability and remission duration of UVA 1 therapy versus 5-MOP UVA photochemotherapy for patients with severe generalized atopic dermatitis.

DETAILED DESCRIPTION:
The patients will be randomized assigned to UVA 1 phototherapy or to 5-MOP UVA photochemotherapy as a first therapy. Besides emollients no additional treatment will be allowed. First a detailed history inclusive drug history will be gathered. The skin type will be determined and a clinical photo will be made. Prior to 5-MOP UVA photochemotherapy an ophthalmological examination, blood cell count and blood chemistry will be routinely performed. A determination of the serum level of 5 MOP will be routinely made at the minimal phototoxic dose (MPD) determination before start of the 5-MOP UVA photochemotherapy. The serum levels of total Ig E and eosinophilic cationic protein (ECP) will be additionally determined at the start and at the end of each therapy. In all patients receiving 5-MOP UVA photochemotherapy reliable eye protection by wearing photoprotective glasses during the treatment and on the day of taking 5-MOP until night will take place. The skin of the patients should not be exposed to direct sun light or to other artificial UV sources at the day of irradiation. A determination of SCORAD Score will be performed by a blinded investigator at baseline, after 10 and 15 irradiations as well as at every follow-up visit at month 1, 3, 6 and 12. A clinical photo will be made at the beginning of each therapy, at the end as well as at every follow-up visit. In case of a relapse (SCORAD Score > 50 % of initial value), or on patients' request for a premature resumption of the therapy (despite SCORAD Score > 50 %) patients will receive that treatment which have not been performed until now. That means, patients who were treated with 5-MOP UVA as a first therapy will now receive the UVA 1 phototherapy and vice versa. The minimum interval between the two therapies is at least 1 month except in a case of complete non response on the first therapy.

Irradiation protocol of the UVA 1 phototherapy:

Irradiation 5 x week for 3 weeks (altogether 15 exposures) Determination of the UVA 1 MED prior to treatment Start with 1 MED if MED < 70 J/cm2. Increase of the dose by 20 % every time if there is not an erythematous reaction and by good tolerability until a maximal dose of 70 J/cm2.

Irradiation protocol of the 5-MOP UVA photochemotherapy:

Irradiation 3 x week for 5 weeks (altogether 15 exposures) Intake of 5-methoxypsoralen (Geralen) 2 hours prior to each irradiation in a dose of 1.2 mg/kg Determination of a minimal phototoxic dose (MPD) prior to treatment Determination of the 5-MOP serum level at the MPD testing Start with 70 % of MPD, no dose increments during the first week. From the second week increase of the UVA dose by 20 % if there is no an erythematous response (respectively by 10 % if there is a light erythemal reaction), but at the earliest 96 hours after the last increment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe generalized atopic dermatitis (SCORAD Score > 45)
* Patients older than 18 years

Exclusion Criteria:

* SCORAD Score < 45
* Pregnant and lactating women
* Patients with severe general diseases
* Abnormal UVA sensitivity
* Intake of photosensitizing drugs
* Local corticosteroid treatment < 2 weeks before entering the study
* Photo(chemo)therapy or systemic treatment for atopic dermatitis < 4 weeks before the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
remission duration after UVA1 phototherapy and after 5-MOP UVA photochemotherapy | 12 months

SECONDARY OUTCOMES:
SCORAD Score at the end of therapy and at 1,3,6 and 12 months after therapy; total IgE and ECP values at the beginning and the end of therapy; cumulative UVA doses; side effects | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Tanew, Prof. MD, Principal Investigator — Medical University of Vienna; University Clinic of Dermatology; Division of Special and Environmental Dermatology
Locations (1):
- Medical University of Vienna; University Clinic of Dermatology; Division of Special and Environmental Dermatology, Vienna, Vienna, Austria